CLINICAL TRIAL: NCT07284589
Title: Evaluation of Ultralow Dose PET Imaging for Detecting SSTR2 Radiotracer Uptake
Brief Title: Ultralow Dose PET Imaging of SSTR2 Radiotracer Uptake
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akiva Mintz (Other)
Responsible Party: Sponsor-Investigator, Akiva Mintz, Executive Director, Nuclear Imaging Institute
Organization: Nuclear Imaging Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NII-0008-SSTR
Record Dates: First submitted 2025-12-08; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy (Controls); Healthy Volunteers; Neuroendocrine (NE) Tumors
Keywords: PET; PET/CT; SSTR2; neuroendocrine; dotatate; low dose; nuclear imaging
MeSH Terms: conditions — Neoplasms | interventions — gallium Ga 68 dotatate; Magnetic Resonance Spectroscopy; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, single-center imaging study designed to evaluate the optimal timing and reconstruction parameters for ultralow dose PET imaging using a long axial field-of-view (LAFOV) PET scanner.
  The study aims to determine whether normal and diseased tissue can be accurately visualized at significantly lower radiotracer doses, while optimizing scan duration and reconstruction methods to maintain diagnostic performance.
  A total of 200 participants will be enrolled in a single cohort, including healthy volunteers and individuals with suspected or confirmed neuroendocrine tumors. The inclusion of both healthy and diseased subjects allows for a comprehensive evaluation of normal organ uptake patterns, which is the primary objective of the study. Participants will undergo a single PET scan session per an enrollment, and be eligible for re-enrollment after 6 months, for a maximum of 5 enrollments if they meet criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ultralow dose 68Ga-DOTATATE imaging group (Other): Participants will be enrolled for an ultralow dose PET scan to evaluate image quality and optimize timing and reconstruction after reducing radiation doses 10-100 fold. Participants will be injected with a very small amount of radiotracer and imaged on a PET scanner for up to 3 hours
  Interventions: Drug: 68Ga-Dotatate

INTERVENTIONS:
Drug: 68Ga-Dotatate — Participants will be injected with 68Ga-DOTATATE and imaged for up to 3 hours on a PET scanner
  Other Names: CT scan; PET scan; blood collection

SUMMARY:
The goal of this clinical trial is to evaluate an investigational ultralow dose positron emission tomography (PET) imaging technique for neuroendocrine tumor detection and monitoring. The main question it aims to answer is:

Can the investigators optimize the timing, scan duration, and image reconstruction to reduce the radiation dose 10-100 fold of the current clinical standard? Participants will be injected with a radioactive tracer that binds to a tumor specific protein called somatostatin receptor 2 (SSTR2) and be imaged on a new type of high sensitivity PET scanner for up to 3 hours

DETAILED DESCRIPTION:
This research study aims to evaluate an investigational ultralow dose PET imaging technique for neuroendocrine tumor detection and monitoring. "Investigational" means that the procedure or drug being studied is not yet approved by the U.S. Food and Drug Administration (FDA) for the specific use being tested in this research. The PET imaging technique used in this study is considered investigational because it is being tested at an ultralow radiation dose that has not yet been approved for clinical use. The radiotracer, Gallium-68 (68Ga)-Dotatate, is FDA-approved for detecting neuroendocrine cancer at standard doses.

68Ga-Dotatate is often found to be taken up at higher levels in in neuroendocrine tumors. In this study, investigators will use a very small amount of this tracer (less than 1/20th of the standard dose) along with advanced PET imaging technology to see if it is possible to create clear images while using much less radiation. This study aims to develop a safer imaging technique that could potentially be used more frequently for screening and treatment response.

Investigators will enroll individuals with and without neuroendocrine tumors to evaluate how ultralow dose PET imaging detects radiotracer uptake in different type of tissue.

Approximately 200 people will be enrolled in this study at the Nuclear Imaging Institute.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Ability to provide informed consent and comply with study procedures.
* For female participants: Must not be pregnant or breastfeeding; Negative pregnancy test required for women of childbearing potential.

Exclusion Criteria:

* Participants who have exceeded NRC regulation for annual radiation exposure from prior research-related scans, including this study (50 millisievert [mSv] total).
* More than four prior enrollments in this study.
* Participants with severe claustrophobia, chronic pain, or musculoskeletal conditions that prevent completion of the PET scan
* Medication & Prior Treatment Exclusions: SSTR targeted therapies
* Pregnant or breastfeeding individuals (negative pregnancy test required)
* Inability to provide informed consent
* Any condition that, in the investigator's judgment, may compromise participant safety or study integrity.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Signal-to-Noise Ratio (SNR) | Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Measurement of signal-to-noise ratio for image quality assessment across different scan durations, reconstruction techniques, and artificial intelligence (AI)-enhanced image reconstructions.
  Unit of Measure: SNR (unitless, numeric ratio)
Contrast-to-Noise Ratio (CNR) | Time Frame: Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Measurement of contrast-to-noise ratio for image quality assessment across different scan durations, reconstruction techniques, and AI-enhanced image reconstructions.
  Unit of Measure: CNR (unitless, numeric ratio)
Coefficient of Variation (COV) | Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Measurement of the coefficient of variation in selected regions for evaluating image consistency across different scan durations, reconstruction techniques, and AI-enhanced image reconstructions.
  Unit of Measure: Percentage (%)
Spatial Resolution (Full Width at Half Maximum - FWHM) | Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Assessment of spatial resolution using full width at half maximum (FWHM) across different scan durations, reconstruction techniques, and AI-enhanced image reconstructions.
  Unit of Measure: Millimeters (mm)
Target-to-Background Ratio (TBR) | Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Assessment of target-to-background ratio for evaluating SSTR2-expressing tissue contrast across different scan durations, reconstruction techniques, and AI-enhanced image reconstructions.
  Unit of Measure: Ratio (unitless numeric ratio)
Qualitative Image Quality Score (Likert Scale) | Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Independent qualitative evaluation of overall image quality, lesion detectability, image noise, and artifacts by nuclear medicine physicians, assessed using a 5-point Likert scale.
  Unit of Measure: Score on Likert Scale (1-5; 1 = worst, 5 = best)
Inter-reader Agreement (Weighted Kappa Statistics) | Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Measurement of agreement among readers evaluating qualitative image quality scores, analyzed using weighted kappa statistics.
  Unit of Measure: Weighted kappa statistic (numeric value ranging from 0 to 1, 0 = no agreement, 1 = perfect agreement)

CONTACTS AND LOCATIONS:
Locations (1):
- Nuclear Imaging Institute, Englewood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
IDP sharing status is currently undecided pending internal review.